CLINICAL TRIAL: NCT02621047
Title: The Effect of Hepatic Impairment on the Pharmacokinetics of Alectinib: A Multiple-Center, Open-Label Study Following Single Oral Dosing of Alectinib to Subjects With Hepatic Impairment and Matched Healthy Subjects With Normal Hepatic Function
Brief Title: Effect of Hepatic Impairment on the Pharmacokinetics of Alectinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP29783; 2015-002976-25 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-11

CONDITIONS: Hepatic Impairment
Keywords: Healthy volunteer; Alectinib; Hepatic impairment
MeSH Terms: interventions — alectinib

ARMS (3):
- Alectinib: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (based on Child-Pugh score) will receive alectinib at a single oral dose of 300 milligrams (mg) on Day 1.
  Interventions: Drug: Alectinib
- Alectinib: Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (based on Child-Pugh score) will receive alectinib at a single oral dose of 300 mg on Day 1.
  Interventions: Drug: Alectinib
- Alectinib: Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive alectinib at a single oral dose of 300 mg on Day 1.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive alectinib as per the dosage schedule mentioned in arm description.

SUMMARY:
This is a multicenter, non-randomized, single-dose, open-label study conducted in male and surgically sterile or post-menopausal female participants with stable chronic hepatic impairment and in healthy participants matched by age, gender, and body weight to assess the effect of hepatic impairment on the pharmacokinetics of alectinib.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Body mass index between 18 to 35 kilograms per square meter (kg/m^2) inclusive and weight greater than (>) 50 kilograms (kg)
* Female participants must be surgically sterile or post-menopausal
* Male participants and their partners of child-bearing potential must be willing to use 2 effective methods of contraception, one of which must be a barrier method

Participants with Hepatic Impairment

- Documented chronic stable liver disease (Child-Pugh Class A, B or C)

Exclusion Criteria:

All Participants

* Pregnant or lactating women, males with female partners who are pregnant or lactating, or women of child bearing potential
* Positive test for drugs of abuse or alcohol
* Participation in an investigational drug or device study within 45 days or 5 half-lives (whichever time period is longer) or 6 months for biologic therapies prior to study drug administration
* History of hypersensitivity to any of the additives in the alectinib formulation
* Participants under judicial supervision, guardianship, or curatorship
* History of severe drug-related allergic reactions or drug-induced hepatotoxicity

Healthy Participants

* Use of any medications (prescription or over-the-counter), within 2 weeks or 5 half-lives (whichever longer) prior to study drug administration
* Use of any herbal supplements or any metabolic inducers within 4 weeks, or 5 half-lives (whichever is longer) prior to study drug administration

Participants with Hepatic Impairment

* Positive screening test for human immunodeficiency virus (HIV)
* History of liver transplantation
* Hepatocellular carcinoma or acute liver disease
* Severe ascites at screening or admission to the clinic
* Recent history (past 2 years) or current severe hepatic encephalopathy (Grade 3 or higher)
* Any evidence of progressive liver disease within the last 4 weeks
* Presence of surgically created or transjugular intrahepatic portal systemic shunts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Pharmaceutical Research Associates CZ, s.r.o., Prague, Czechia
- Summit Clinical Research s.r.o.; Oddelenie internej mediciny a klinickej farmakologie, Bratislava, Slovakia

REFERENCES:
- [Derived] Morcos PN, Cleary Y, Sturm-Pellanda C, Guerini E, Abt M, Donzelli M, Vazvaei F, Balas B, Parrott N, Yu L. Effect of Hepatic Impairment on the Pharmacokinetics of Alectinib. J Clin Pharmacol. 2018 Dec;58(12):1618-1628. doi: 10.1002/jcph.1286. Epub 2018 Jul 27. PMID 30052269

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 'Alectinib: Normal Hepatic Function' participants were grouped into 2 arms: 'Alectinib: Normal Moderate Matched Control' and 'Alectinib: Normal Severe Matched Control'. Same 'Alectinib: Normal Hepatic Function' participant could be included in both 'Alectinib: Normal Moderate Matched Control' and 'Alectinib: Normal Severe Matched Control' arms.
Groups:
- Alectinib: Moderate Hepatic Impairment: Participants with moderate hepatic impairment (based on Child-Pugh score) received alectinib at a single oral dose of 300 milligrams (mg) on Day 1.
- Alectinib: Severe Hepatic Impairment: Participants with severe hepatic impairment (based on Child-Pugh score) received alectinib at a single oral dose of 300 mg on Day 1.
- Alectinib: Normal Hepatic Function: Participants with normal hepatic function received alectinib at a single oral dose of 300 mg on Day 1.
Period: Overall Study
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Hepatic Function
Started | 8 | 8 | 12
Completed | 8 | 8 | 11
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled in the study and received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 8 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (8.52) | 53.1 (5.62) | 52.2 (7.98) | 53.1 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 12
  Male | 5 | 4 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins
Time Frame: Predose (0 hour), and at 1, 2, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, and 240 hours postdose (Dosing day = Day 1)
Population: Pharmacokinetic population included all participants who were enrolled in the study, received study treatment, and had pharmacokinetic data available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Alectinib: Normal Moderate Matched Control: Participants with normal hepatic function matched to the participants in moderate hepatic impairment group (based on Child-Pugh score), on the basis of age, body weight and gender, received alectinib at a single oral dose of 300 mg on Day 1.
- Alectinib: Normal Severe Matched Control: Participants with normal hepatic function matched to the participants in severe hepatic impairment group (based on Child-Pugh score), on the basis of age, body weight and gender, received alectinib at a single oral dose of 300 mg on Day 1.
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanograms per milliliter (ng/mL) | 107 (35.9) | 83.6 (58.4) | 85.5 (54.4) | 85.1 (85.0)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio Percentage (%) = 128, 90% CI 2-sided [86.5 to 188]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 100, 90% CI 2-sided [55.1 to 183]

2. Primary Outcome: Cmax of Unbound Alectinib
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 24.0 (35.3) | 16.2 (38.7) | 16.1 (33.1) | 12.3 (87.0)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 148, 90% CI 2-sided [106 to 208]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 130, 90% CI 2-sided [75.4 to 225]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC 0-inf) for Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins. AUC 0-inf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC 0-t plus AUC t-inf.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 2920 (60.5) | 1830 (40.4) | 3850 (54.1) | 1750 (64.0)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 160, 90% CI [105 to 243]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 220, 90% CI [131 to 369]

4. Primary Outcome: AUC 0-inf for Unbound Alectinib
Description: AUC 0-inf = AUC from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC 0-t plus AUC t-inf.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 659 (60.5) | 355 (27.4) | 725 (37.8) | 254 (70.6)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 186, 90% CI [122 to 281]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 285, 90% CI [175 to 466]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measureable Concentration (AUC 0-last) for Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 2820 (63.7) | 1740 (45.1) | 3710 (56.6) | 1630 (74.8)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 162, 90% CI 2-sided [104 to 254]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 228, 90% CI [129 to 403]

6. Primary Outcome: AUC 0-last for Unbound Alectinib
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 636 (63.3) | 337 (31.9) | 699 (38.9) | 236 (80.2)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 189, 90% CI [121 to 293]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 296, 90% CI 2-sided [174 to 506]

7. Secondary Outcome: Cmax of Total Metabolite of Alectinib (M4)
Description: Total M4 = unbound M4 plus M4 bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 19.3 (62.0) | 29.8 (89.3) | 17.5 (114) | 28.7 (99.5)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 64.6, 90% CI [36.2 to 115]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 60.8, 90% CI 2-sided [26.6 to 139]

8. Secondary Outcome: Cmax of Unbound M4
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 17.6 (51.3) | 20.6 (45.4) | 8.26 (39.6) | 14.0 (82.7)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 85.1, 90% CI [55.5 to 130]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 59.0, 90% CI [34.2 to 102]

9. Secondary Outcome: Cmax of Total Combined Alectinib and M4 (Alectinib + M4)
Description: Total alectinib + M4 = unbound alectinib + M4 plus alectinib + M4 bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanomoles per liter (nmol/L) | 266 (23.3) | 229 (65.6) | 214 (61.3) | 218 (90.5)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 116, 90% CI [78.6 to 172]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 98.1, 90% CI [51.7 to 186]

10. Secondary Outcome: Cmax of Unbound Alectinib + M4
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
nmol/L | 87.0 (24.4) | 75.9 (39.5) | 48.9 (36.1) | 50.6 (86.4)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 115, 90% CI 2-sided [85.2 to 154]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 96.6, 90% CI 2-sided [55.6 to 168]

11. Secondary Outcome: AUC 0-inf of Total M4
Description: Total M4 = unbound M4 plus M4 bound to plasma proteins. AUC 0-inf = AUC from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC 0-t plus AUC t-inf.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 583 (14.8) | 718 (70.5) | 465 (147) | 709 (92.4)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 80.6, 90% CI [50.2 to 130]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 65.6, 90% CI 2-sided [26.9 to 160]

12. Secondary Outcome: AUC 0-inf of Unbound M4
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 516 (27.3) | 497 (33.7) | 220 (71.1) | 345 (77.8)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 104, 90% CI [76.8 to 141]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 63.7, 90% CI 2-sided [34.0 to 119]

13. Secondary Outcome: AUC 0-inf of Total Alectinib + M4
Description: Total alectinib + M4 = unbound alectinib + M4 plus alectinib + M4 bound to plasma proteins. AUC 0-inf = AUC from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC 0-t plus AUC t-inf.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nmol/L
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nmol/L | 7340 (46.6) | 5380 (44.5) | 9020 (60.3) | 5120 (74.9)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 136, 90% CI 2-sided [94.7 to 196]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 176, 90% CI [98.4 to 315]

14. Secondary Outcome: AUC 0-inf of Unbound Alectinib + M4
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nmol/L
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nmol/L | 2420 (38.5) | 1800 (25.4) | 1960 (41.3) | 1250 (78.7)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 134, 90% CI [99.6 to 181]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 157, 90% CI 2-sided [91.8 to 268]

15. Secondary Outcome: AUC 0-last of Total M4
Description: Total M4 = unbound M4 plus M4 bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 475 (27.5) | 648 (79.6) | 363 (212) | 631 (109)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 73.3, 90% CI 2-sided [46.2 to 116]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 57.5, 90% CI 2-sided [20.0 to 165]

16. Secondary Outcome: AUC 0-last of Unbound M4
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*ng/mL | 433 (29.6) | 448 (40.2) | 172 (100) | 308 (90.8)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 96.6, 90% CI [69.9 to 134]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 55.8, 90% CI [26.0 to 120]

17. Secondary Outcome: AUC 0-last of Total Alectinib + M4
Description: Total alectinib + M4 = unbound alectinib + M4 plus alectinib + M4 bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nmol/L
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nmol/L | 7160 (47.6) | 5170 (48.2) | 8700 (62.7) | 4830 (82.4)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 139, 90% CI 2-sided [94.8 to 203]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 180, 90% CI [97.2 to 334]

18. Secondary Outcome: AUC 0-last of Unbound Alectinib + M4
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nmol/L
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nmol/L | 2390 (38.4) | 1750 (27.5) | 1890 (42.7) | 1200 (81.1)
Statistical Analysis 1: Comparison: Alectinib: Moderate Hepatic Impairment vs Alectinib: Normal Moderate Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 137, 90% CI 2-sided [100 to 186]
Statistical Analysis 2: Comparison: Alectinib: Severe Hepatic Impairment vs Alectinib: Normal Severe Matched Control; Test type: Superiority or Other; Geometric Mean Ratio % = 158, 90% CI 2-sided [91.2 to 274]

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: hours
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 6.04 [3.82 to 23.8] | 5.97 [3.98 to 6.10] | 7.02 [2.00 to 11.9] | 4.97 [3.90 to 6.10]

20. Secondary Outcome: Tmax for Total M4
Description: Total M4 = unbound M4 plus M4 bound to plasma proteins
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: hours
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 8.10 [6.07 to 35.8] | 7.88 [5.92 to 10.0] | 8.00 [5.98 to 11.9] | 8.05 [5.93 to 11.6]

21. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins. t1/2 = the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 26.1 (26.1) | 20.1 (21.1) | 39.3 (27.0) | 22.2 (31.5)

22. Secondary Outcome: t1/2 of Total M4
Description: Total M4 = unbound M4 plus M4 bound to plasma proteins. t1/2 = the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 24.5 (48.0) | 19.3 (18.0) | 30.5 (68.8) | 20.1 (30.4)

23. Secondary Outcome: Apparent Oral Clearance (CL/F) of Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins. Clearance is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the oral bioavailability.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
liters per hour | 103 (60.5) | 164 (40.4) | 77.9 (54.1) | 171 (64.0)

24. Secondary Outcome: CL/F of Unbound Alectinib
Description: Clearance is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the oral bioavailability.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
liters per hour | 455 (60.5) | 845 (27.4) | 414 (37.8) | 1180 (70.6)

25. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins. Volume of distribution is defined as the theoretical volume which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose is influenced by the fraction absorbed.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
liters | 3870 (55.7) | 4760 (61.3) | 4410 (73.0) | 5490 (86.5)

26. Secondary Outcome: Vz/F for Unbound Alectinib
Description: Volume of distribution is defined as the theoretical volume which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose is influenced by the fraction absorbed.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
liters | 17200 (51.8) | 24500 (47.0) | 23400 (52.7) | 37800 (95.6)

27. Secondary Outcome: Fraction of Drug Unbound (fu) of Total Alectinib
Description: Total alectinib = unbound alectinib plus alectinib bound to plasma proteins. fu = ratio of unbound alectinib to total alectinib multiplied by 100.
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of total alectinib
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Normal Moderate Matched Control | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Severe Matched Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
percentage of total alectinib | 0.225 (18.3) | 0.194 (28.4) | 0.188 (37.8) | 0.145 (36.7)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 21
Description: Safety population
Arm/Group | Alectinib: Moderate Hepatic Impairment | Alectinib: Severe Hepatic Impairment | Alectinib: Normal Hepatic Function
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/12
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib: Moderate Hepatic Impairment (N=8) | Alectinib: Severe Hepatic Impairment (N=8) | Alectinib: Normal Hepatic Function (N=12)
Angina unstable (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib: Moderate Hepatic Impairment (N=8) | Alectinib: Severe Hepatic Impairment (N=8) | Alectinib: Normal Hepatic Function (N=12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.